CLINICAL TRIAL: NCT05675696
Title: Assessment of Occult Lung Stress During Lung Protective Mechanical Ventilation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The company that was providing the catheters lost funding, and the study will not be moving forward.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-00695
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ARDS Patients Intubated on Mechanical Ventilation (Experimental): ARDS patients in the ICU who are intubated on mechanical ventilation will be included. During ventilation, an esophageal catheter will be used to measure the esophageal pressure, which estimates pleural pressure at the level of the catheter. The esophageal catheter's position will be confirmed by a chest radiograph once inserted. The ventilator settings may be changed to see if these ventilator adjustments can reduce potential lung stress in ARDS patients. There is no set criteria for adjusting the ventilator settings based on the study device, but the goal would be to adjust the volume until the inspiratory effort measured by the catheter disappears so as to protect the patient. A one-to-two-hour study session will be performed for data collection. The esophageal catheter will be removed at the end of the study session or can be left in place for use as a feeding tube if needed for patient care.
  Interventions: Other: Esophageal Catheter

INTERVENTIONS:
Other: Esophageal Catheter — Newly designed external monitor that will capture esophageal pressure from a proprietary nasogastric tube combined with simultaneous pressure, flow, and volume measurements from the ventilator tubing.
  Other Names: PulmoTech Esophageal Pressure System (iEPS)

SUMMARY:
The present study will utilize esophageal manometry to measure the presence and magnitude of persistent patient effort during lung protective ventilation, allowing identification and mitigation of occult lung stress.

ELIGIBILITY:
Inclusion Criteria:

* Intubated with a diagnosis of ARDS and expected to be ventilated for ≥ 48 hours
* Meets Berlin criteria for ARDS, with or without underlying chronic lung disease
* Triggering breaths on the ventilator
* Treating medical team agrees with patient participation

Exclusion Criteria:

* Known or suspected esophageal abnormalities, craniofacial abnormalities, or upper GI bleed
* Shock that requires ≥ 2 vasopressors
* pH on arterial blood gas ≤7.25
* Minute ventilation ≥ 14L/min
* Known or suspected pneumothorax, pneumomediastinum, and/or subcutaneous emphysema
* Severe ARDS with P/F ratio <60
* Pregnancy
* Currently receiving extracorporeal membrane oxygenation (ECMO) therapy
* Decision to withhold life-sustaining treatment
* Patients who are not expected to survive for 24 hours
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Transpulmonary Driving Pressure | Up to Hour 2 (Day 1)
  Transpulmonary driving pressure is the pressure difference between the airway opening and pleural surface. It represents lung stress and is higher with increased spontaneous respiration and work of breathing.
Driving Pressure | Up to Hour 2 (Day 1)
  Driving pressure is defined as plateau pressure minus positive end-expiratory pressure (PEEP). Driving pressure during mechanical ventilation is directly related to stress forces in the lung.
Work of Breathing (WOB) | Up to Hour 2 (Day 1)
  WOB is the amount of energy or oxygen (O2) consumption needed by the respiratory muscles to produce enough ventilation and respiration to meet the metabolic demands of the body.
Pressure-Time Product (PTP) | Up to Hour 2 (Day 1)
  PTP is the product of the average inspiratory pressure (starting from the onset of effort) and the duration of inspiration. The PTP was developed to account for energy expenditures during the dynamic and isometric phases of respiration.

SECONDARY OUTCOMES:
Lung Compliance (C, l) | Up to Hour 2 (Day 1)
  Lung compliance is calculated as the tidal volume divided by the difference of transpulmonary pressure at end inspiration minus transpulmonary pressure at PEEP:
  (C, l) = tidal volume/(transpulmonary pressure at end inspiration - transpulmonary pressure at PEEP).
  Expressed in (ml/cmH2O).
Chest Wall Compliance (C, cw) | Up to Hour 2 (Day 1)
  Chest wall compliance is calculated as the tidal volume divided by the difference of esophageal pressure at end inspiration minus esophageal pressure at PEEP:
  (C, cw) = tidal volume/(esophageal pressure at end inspiration - esophageal pressure at PEEP).
  Expressed in (ml/cmH2O).
Respiratory System Compliance (C, rs) | Up to Hour 2 (Day 1)
  Respiratory System Compliance is calculated as the tidal volume divided by the difference of the airway pressure at end inspiration minus airway pressure at PEEP:
  (C, rs) = tidal volume/(airway pressure at end inspiration - airway pressure at PEEP).
  Expressed in (ml/cmH2O).
Oxygen Saturation | Up to Hour 2 (Day 1)
  Oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin in the blood.
PaO2/FiO2 (P/F) Ratio | Up to Hour 2 (Day 1)
  The P/F ratio is the arterial partial pressure of oxygen (PaO2) divided by the inspired oxygen concentration (FiO2).

CONTACTS AND LOCATIONS:
Overall Officials: Beno Oppenheimer, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- Tisch Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Beno Oppenheimer [Beno.Oppenheimer@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposes to use the data will be granted access upon reasonable request. Requests should be directed to Beno.Oppenheimer@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.